CLINICAL TRIAL: NCT01902355
Title: Comparison of Two Needle Insertion Techniques on Success Rate and Complications During Central Venous Catheterization: Seldinger vs. Modified Seldinger Technique
Brief Title: Comparison of Two Needle Insertion Techniques on Success Rate and Complications During Central Venous Catheterization
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Deok Man Hong, Assistant Professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: modifiedSeldinger; H1305617491 (Other: SNUH)
Record Dates: First submitted 2013-07-15; First posted 2013-07-18 (Estimated); Last update posted 2014-07-03 (Estimated); Status verified 2014-07

CONDITIONS: Complications of Central Venous Catheterization
Keywords: Central Venous Catheterization

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- modified Seldinger technique (Experimental): Use needle that is covered with guiding sheath. After desired vessel puncture, guiding sheath is instantly slid over the needle into the vessel. The needle is withdrawn, guidewire is advanced through the guiding sheath, central catheter is placed into the vessel.
  Interventions: Procedure: modified Seldinger technique
- Seldinger technique (Active Comparator): The desired vessel is punctured with a sharp hollow needle, syringe is detached and guidewire is advanced through the lumen of the needle, and then the needle is withdrawn. Central catheter is then passed over the guidewire into the vessel.
  Interventions: Procedure: Seldinger technique

INTERVENTIONS:
Procedure: modified Seldinger technique — modified Seldinger technique(guiding sheath-over-the-needle technique) use needle that is covered with guiding sheath. After desired vessel puncture, guiding sheath is instantly slid over the needle into the vessel. The needle is withdrawn, guidewire is advanced through the guiding sheath, central catheter is placed into the vessel.
  Arms: modified Seldinger technique
Procedure: Seldinger technique — The desired vessel is punctured with a sharp hollow needle, syringe is detached and guidewire is advanced through the lumen of the needle, and then the needle is withdrawn. Central catheter is then passed over the guidewire into the vessel.
  Arms: Seldinger technique

SUMMARY:
The purpose of this study is to compare two needle insertion techniques(Seldinger vs. modified Seldinger technique) on success rate and complications during central venous catheterization.

DETAILED DESCRIPTION:
Unintended arterial puncture and local hematoma formation are the most common complications during internal jugular vein central venous catheterization. Other serious complications like pseudoaneurysm, arteriovenous fistula, arterial dissection, thrombosis, embolism are also possible. These complications mostly occur by mechanical trauma or injury when advancing needle back and forth to puncture internal jugular vein. Placement of guidewire or dilator can also cause mechanical trauma or injury around the vessel.

Because internal jugular vein collapses easily during needle advance, anterior and posterior wall of the vessel can be punctured simultaneously. Posterior wall puncture can increase the risk of complications of the catheterization. Delicate puncture of the vessel and stable fixation of the needle after puncture are important to reduce overall number of catheterization attempts, increase success rate, reduce complications.

Seldinger technique(thin-wall needle technique) is commonly used procedure to obtain safe access to central vein. The desired vessel is punctured with a sharp hollow needle, syringe is detached and guidewire is advanced through the lumen of the needle, and then the needle is withdrawn. Central catheter is then passed over the guidewire into the vessel. Contrarily, modified Seldinger technique(guiding sheath-over-the-needle technique) use needle that is covered with guiding sheath. After desired vessel puncture, guiding sheath is instantly slid over the needle into the vessel. The needle is withdrawn, guidewire is advanced through the guiding sheath, central catheter is placed into the vessel.

When using Seldinger technique, it is important to fix the needle firmly with hand until the guidewire is placed into the vessel lumen. If hand fixation is not stable, needle tip can migrate from the lumen, can pierce the vessel wall, and carotid artery puncture, and local hematoma formation might occur. Even if there is no evidence of complications, when blood regurgitation fails, overall number of vessel puncture attempts would increase and it is expected that rate of complications of the catheterization would increase.

When using modified Seldinger technique, guiding sheath is easily slid over the needle, providing stable route into the vessel lumen relatively in early step of the catheterization. Therefore, it is expected that stability of the fixation improves, success rate of the catheterization increase, and complications of the catheterization decrease. But there is no high level of evidence yet, and still decision to use which technique is based on experience of the operator.

Investigators are going to compare the Seldinger technique and modified Seldinger technique on success rate and complications during central venous catheterization by prospective, randomized, controlled study.

ELIGIBILITY:
Inclusion Criteria:

* patient scheduled for surgery and internal jugular vein central catheterization

Exclusion Criteria:

* Patient who doesn't agree to the study
* Catheterization site inflammation
* Contralateral diaphragmatic dysfunction
* Anatomic anomalies of carotid artery or vein
* Previous neck surgical history
* Recent(less than 1 month) right internal jugular vein central catheterization

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 272 (Actual)
Dates: Start 2013-07; Primary Completion 2014-06 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
number of attempts of guidewire advance | after internal jugular vein puncture
  after desired vessel is punctured guidewire is advanced through the lumen of the needle or guiding sheath

SECONDARY OUTCOMES:
complications of internal jugular vein central catheterization | after central catheter placement
  any complications including arterial puncture, hematoma of skin and subcutaneous tissue, pneumothorax, hemothorax
  - evaluate with ultrasonography and compare with pre-catheterization image

CONTACTS AND LOCATIONS:
Overall Officials: Deok Man Hong, M.D., Ph. D., Study Chair — Seoul National University Hospital; Tae Kyong Kim, M.D., Study Director — Seoul National University of Hospital
Locations (1):
- Seoul National University of Hospital, Seoul, South Korea